CLINICAL TRIAL: NCT00651105
Title: A Double-blind, Placebo-controlled, Randomized, Cross-over Study to Evaluate the GLP-1-mediated and Non-GLP-1-mediated Effects of LAF237 on Glucagon Secretion in Patients With Type 2 Diabetes and in Healthy Subjects
Brief Title: Effect of LAF237 on Glucagon Secretion in Patients With Type 2 Diabetes and in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2347
Record Dates: First submitted 2008-03-28; First posted 2008-04-02 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Type-2 Diabetes; Healthy
Keywords: Diabetes; Hyperglycemia; Healthy; Vildagliptin; Adults
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Vildagliptin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to assess the GLP-1 and non-GLP-1 effects of LAF237 on glucagon secretion, using treatment observations of the overall glycemic response.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria - Type-2 Diabetes Patients

* Male or female patients aged 30 to 75 years with Type-2 Diabetes Mellitus (T2DM) and who are in otherwise good health
* Must have been diagnosed with T2DM at least 6 months prior to screening, and whose diabetes is controlled by diet and exercise alone or by stable dosage ( > 3 months) of metformin
* HbA1c in the range of 6.5% to 9% at screening

Inclusion Criteria - Healthy Volunteers

* Male or female subjects aged 30 to 75 years, determined to be in good health
* Normal oral glucose tolerance test (OGTT) at screening
* Age, gender and weight matched to subjects with T2DM

Exclusion Criteria:

Exclusion criteria - Type-2 Diabetes Patients

* A history of:
* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g., Cushing's syndrome and acromegaly
* Acute metabolic diabetic complications (such as ketoacidosis or hyperosmolar state (coma)) within the past 6 months
* Torsades de Pointes, ventricular tachycardia or ventricular fibrillation
* Any severe hypoglycemic episode within 3 months of screening
* Use of any of the following medications:
* Antihypertensive or lipid-lowering agents unless on a stable dose for at least 3 months prior to screening
* Chronic insulin treatment (> 4 weeks of treatment in the absence of an intercurrent illness) within the past 6 months
* Chronic oral/intramuscular/intravenous corticosteroid treatment ( > 7 consecutive days of treatment) within 8 weeks prior to screening

Exclusion Criteria - Healthy Volunteers

* First degree relative of an individual with T2DM
* History of gestational diabetes
* Use of any prescription medication within 1 month prior to dosing. Use of over-the-counter medications or vitamins within 14 days prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
GLP-1 and non GLP-1 effects of LAF237 on glucagon secretion in patients with Type-2 diabetes and matching healthy subjects | from baseline to Day 10

SECONDARY OUTCOMES:
Effects of LAF237 on prandial glucose profiles, prandial insulin, and gastric-emptying in patients with Type-2 diabetes and in matching healthy subjects. | 10 day treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (2):
- Germany (2):
  - Novartis Investigator Site, Bad Lauterberg im Harz
  - Novartis Investigator Site, Berlin

REFERENCES:
- [Result] Nauck MA, Kind J, Kothe LD, Holst JJ, Deacon CF, Broschag M, He YL, Kjems L, Foley J. Quantification of the Contribution of GLP-1 to Mediating Insulinotropic Effects of DPP-4 Inhibition With Vildagliptin in Healthy Subjects and Patients With Type 2 Diabetes Using Exendin [9-39] as a GLP-1 Receptor Antagonist. Diabetes. 2016 Aug;65(8):2440-7. doi: 10.2337/db16-0107. Epub 2016 Apr 5. PMID 27207543